CLINICAL TRIAL: NCT02354144
Title: A Randomized Controlled Trial of a Carrageenan-Containing Lubricant to Reduce Transmission of Human Papillomavirus Infection Among Men Who Have Sex With Men
Brief Title: Lubricant Investigation in Men to Inhibit Transmission of HPV Infection
Acronym: LIMIT-HPV
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Mandated by DSMB
Sponsor: McGill University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dr. Eduardo Franco, James McGill Professor and Chair (Department of Oncology) and Director (Division of Cancer Epidemiology), McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A10-M98-14B; CIHR-MOP-137066 (Other Grant/Funding Number: Canadian Institutes of Health Research); CCSRI-703032 (Other Grant/Funding Number: Canadian Cancer Society Research Institute)
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Human Papillomavirus Infection
Keywords: Human papillomavirus; Carrageenan; Microbicide; Anal HPV infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Carrageenan-containing gel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carrageenan-based gel (Experimental): The intervention to be administered is:
  * a commercially available gel that contains carrageenan.
  * water-based, latex-condom compatible, clear, odourless, tasteless, and have similar viscosity as the placebo gel.
  * also packaged in a similar plastic bottle with a disk cap that can be operated with one finger, and must be applied prior to anal intercourse during the entire study period. Around 15 ml of the personal lubricant will be dispensed into the hand and applied directly to the genital, anal, and condom surfaces prior to and as needed during anal sex. When sexual activity ceases, the water-based formulation of the gel allows it to be easily removed with lukewarm water.
  Interventions: Other: Carrageenan-based gel
- Control gel (Placebo Comparator): The intervention to be administered is:
  * a commercially available gel that does not contain carrageenan.
  * water-based, latex-condom compatible, clear, odourless, tasteless, and have similar viscosity as the carrageenan-containing gel.
  * also packaged in a similar plastic bottle with a disk cap that can be operated with one finger, and must be applied prior to anal intercourse during the entire study period. Around 15 ml of the personal lubricant will be dispensed into the hand and applied directly to the genital, anal, and condom surfaces prior to and as needed during anal sex. When sexual activity ceases, the water-based formulation of the gel allows it to be easily removed with lukewarm water.
  Interventions: Other: Control gel

INTERVENTIONS:
Other: Carrageenan-based gel — Carrageenan is a non-toxic gelling agent safe in animals and humans as a potent HPV inhibitor. An anionic polymer derived from red algae, carrageenan has a long history of human use as a stabilizer and emulsifier in many industries. All three major classes of carrageenan act as extremely potent HPV inhibitors and block HPV infection by binding to the viral capsid, thus preventing attachment to the appropriate cell-surface heparan sulfate proteoglycans (HSPG) receptors.
  Arms: Carrageenan-based gel
Other: Control gel — A gel not containing carrageenan
  Arms: Control gel

SUMMARY:
The LIMIT-Study is a placebo-controlled, double-blinded randomized controlled trial designed to explore the efficacy of a carrageenan-based lubricant as a topical microbicide for preventing HPV acquisition. Individuals at high risk for infection (men who have sex with men, or MSM, and especially those with HIV) will be included in the trial. Participants will complete a self-administered baseline questionnaire during the enrollment visit, and follow-up questionnaires during all other six visits. The shorter follow-up questionnaires are intended to evaluate recent sexual behaviours and to corroborate the responses given during the baseline visit. These questionnaires will measure HPV risk factors, compliance, and monitor safety and tolerability of the gels. Between follow-up visits, participants will be asked to log into a secure web module at least once a week to answer questions on daily sexual activities, condom and study gel use, and adverse events. Individuals will be screened for eligibility over the telephone or in person and eligible men will attend an enrollment visit, where the nurse will obtain informed consent and instruct the participant on gel use. They will receive a one month's supply of gel and provide the first specimen. Random number sets will be assigned to the treatment and control gel. Each participant will be assigned an individual code, which will be used to match him to the study arm. Lastly, the nurse will provide details about HPV infection and advice about condom use and sexual health. HPV infection status will be measured using anal specimens at baseline (enrollment/time 0), and at all follow-up clinic visits (1, 2, 3, 6, 9 and 12 months).

DETAILED DESCRIPTION:
Human papillomavirus (HPV) inhibitory compounds might be useful as topical microbicides for blocking the spread of HPV. Recent in-vitro and in-vivo laboratory studies have demonstrated the strong inhibitory properties of carrageenan (an inexpensive gelling agent that is non-toxic and safe in animals and humans) against all HPV types. So far, there has been no clinical trial designed to assess a carrageenan-based personal lubricant as a topical microbicide in the Men who have Sex with Men (MSM) population. Since the introduction of HAART therapy in 1996, there has been a paradoxical effect on the incidence of anal cancer, a disease caused by HPV. Whereas patients would formerly die of some other AIDS-related ailment, men undergoing HAART therapy now have increased longevity, thus allowing diseases with longer natural history such as anal cancer to develop. Low cluster of differentiation 4 (CD4) counts, high HPV incidence and longer duration of infection have contributed to elevating the risk of anal lesions and cancer among MSMs with HIV to nearly 80 times that of the general male population. Although HPV vaccination has been approved for males in Canada, it is exclusively prophylactic, i.e. it will only prevent HPV infection before exposure occurs. But considering that most MSMs will have already been exposed to the vaccine target types, its benefits in this population are limited. Furthermore, current vaccination only protects against two of the 14 oncogenic HPV types.

The primary aim of the study is to evaluate the efficacy of carrageenan in reducing type-specific anal HPV incidence, i.e., in preventing infections by new HPV types in sexually active MSM. Secondary aims are: 1) to evaluate the efficacy of carrageenan in reducing type-specific anal HPV prevalence, i.e., in accelerating clearance of existing infections in sexually active MSM; 2) to compare the efficacy of carrageenan for type-specific prevention and clearance of anal HPV infections among MSM with and without HIV, i.e., to evaluate whether carrageenan is equally effective among these subgroups; and 3) to assess the safety and tolerability of the proposed gel and patient adherence to the intervention, i.e., the parameters important for future clinical use.

To permit verification of the study's objectives with sufficient power at the end of the one-year follow-up period, we propose to recruit 380 subjects (110 HIV+ and 270 HIV-). We will be recruiting subjects living with HIV through 5 HIV/AIDS outpatient clinics in Montreal: Clinique Médicale du Quartier-Latin, Clinique L'Actuel, Clinique OPUS, Unité d'Hospitalisation de Recherche et d'Enseignement sur les Soins du SIDA (UHRESS) of the Centre Hospitalier de L'Université de Montréal (CHUM) and Chronic Viral Illnesses Service of McGill University Health Centre (MUHC). We will advertise at bars, sex and health clubs, in various media, and the abovementioned clinics-with the addition of the McGill University Student Health Services. MSMs with and without HIV will be recruited. For those with HIV, a chart review will be performed at enrollment to collect information on CD4+ count, viral load, HAART status, year of HIV diagnosis, and nadir CD4+ count. HIV testing will also be performed on MSMs without HIV to verify their status.

Volunteer MSMs living in Montreal will be randomized to receive either a) treatment with carrageenan self-applied as an anal microbicide gel, or b) treatment with a placebo gel applied in the same way. Our specific primary aim is to evaluate the efficacy of carrageenan in reducing anal HPV incidence, i.e., in preventing new HPV infections in sexually active MSMs. Additional secondary aims include: to evaluate the efficacy of carrageenan in reducing anal HPV prevalence (i.e., in accelerating clearance of existing infections in sexually active MSMs), to evaluate if there is a difference in the efficacy of carrageenan for prevention and clearance of HPV infections between individuals living with and without HIV, and to evaluate patient adherence as measured by behavioural characteristics assessed by means of questionnaires.

Participants will be randomized to either carrageenan or placebo gels by a variable block randomization algorithm and blinded intervention. Demographics, risk factor, and compliance information will be collected via computerized questionnaires at baseline (enrollment/ time 0), and 1, 2, 3, 6, 9 and 12 months post-enrollment. HPV DNA detection and genotyping of anal samples will be done at the same clinic visits by the PGMY polymerase chain reaction protocol. Measuring the efficacy of the intervention will be done by testing the null hypothesis of no difference in time to HPV infection (i.e., infection with an HPV type not present at baseline) between treatment groups with the log rank test. We will use a Cox proportional hazards regression model to estimate the hazard ratio and 95% confidence intervals of HPV infection for the treatment versus placebo group. We will also use survival analysis techniques to measure clearance of infections with HPV types present at enrollment according to the intervention. Our analyses will be conducted separately according to participant HIV status, and eventually pooled if results are found to be similar between groups. We will perform our analyses according to the intention-to-treat approach (i.e., including all participants who were randomized and received at least one-month's supply of gel), and the according-to-protocol approach (i.e., including only participants who complied with the protocol).

Considering that HPV infection is responsible for 90% of anal cancer cases, as well as for much suffering due to genital warts, the potential for this microbicide-based approach in disease prevention cannot be overemphasized. Our team has extensive experience in studies of HPV epidemiology in Montreal and subject recruitment resources are already in place.

(Full protocol available upon request)

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 or older,
* Men living in Montreal and plan to remain in the city for the next 12 months,
* Men who have had receptive anal sex with one or more men during the previous 3 months and intend to continue being sexually active for the duration of their involvement in the study, irrespective of whether their sexual partner will change,
* Men planning on having receptive anal sex with two or more men, but less than 50 DIFFERENT partners per year
* Men who understands French or English,
* Men willing to follow study instructions and comply with follow-ups for 12 months.

Exclusion Criteria:

* Men must not be receiving treatment for anal or perianal condylomas or anal intraepithelial neoplasia lesions during the trial,
* Men must not have a known allergy or hypersensitivity to any of the ingredients in either gels.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Franco, DrPH, Principal Investigator — McGill University
Locations (1):
- McGill University - Division of Cancer Epidemiology, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Kassam P, El-Zein M, Tota JE, Tellier PP, Coutlee F, de Pokomandy A, Franco EL. HPV vaccination and anal HPV infection in gay, bisexual, and other men who have sex with men. Vaccine. 2025 Jan 25;45:126644. doi: 10.1016/j.vaccine.2024.126644. Epub 2024 Dec 21. PMID 39708517
- [Derived] Laurie C, El-Zein M, Tota J, Khosrow-Khavar F, Tellier PP, Coutlee F, de Pokomandy A, Franco EL; Lubricant Investigation in Men to Inhibit Transmission of Human Papillomavirus Infection (LIMIT-HPV) Study Group. Efficacy of a Carrageenan Gel in Increasing Clearance of Anal Human Papillomavirus Infections in Men: Interim Analysis of a Double-Blind, Randomized Controlled Trial. J Infect Dis. 2023 Feb 1;227(3):402-406. doi: 10.1093/infdis/jiac019. PMID 35090175
- [Derived] Laurie C, El-Zein M, Tota JE, Khosrow-Khavar F, Tellier PP, Coutlee F, de Pokomandy A, Franco EL; LIMIT-HPV study group. Efficacy of a carrageenan gel in preventing anal human papillomavirus (HPV) infection: interim analysis of the Lubricant Investigation in Men to Inhibit Transmission of HPV Infection (LIMIT-HPV) randomised controlled trial. Sex Transm Infect. 2022 Jun;98(4):239-246. doi: 10.1136/sextrans-2021-055009. Epub 2021 Jun 17. PMID 34140405
- [Derived] Laurie C, El-Zein M, Tota J, Tellier PP, Coutlee F, Franco EL, de Pokomandy A; LIMIT-HPV study group. Lubricant Investigation in Men to Inhibit Transmission of HPV Infection (LIMIT-HPV): design and methods for a randomised controlled trial. BMJ Open. 2020 Mar 23;10(3):e035113. doi: 10.1136/bmjopen-2019-035113. PMID 32205376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Recruitment for the LIMIT-HPV trial began in February 2016 at the following sites in Montreal, Canada: McGill University Health Centre, Clinique Médicale Urbaine du Quartier-Latin, Clinique OPUS, and two student health services clinics (McGill and Concordia universities). From September 2018 to March 2020, study visits were completed at McGill University's Division of Cancer Epidemiology's research clinic. 255 of the 258 participants were enrolled and analyzed at the time of interim analysis.
Groups:
- Carrageenan-based Gel: The intervention to be administered is:
  * a commercially available gel that contains carrageenan.
  * water-based, latex-condom compatible, clear, odourless, tasteless, and have similar viscosity as the placebo gel.
  * also packaged in a similar plastic bottle with a disk cap that can be operated with one finger, and must be applied prior to anal intercourse during the entire study period. Around 15 ml of the personal lubricant will be dispensed into the hand and applied directly to the genital, anal, and condom surfaces prior to and as needed during anal sex. When sexual activity ceases, the water-based formulation of the gel allows it to be easily removed with lukewarm water.
  Carrageenan-based gel: Carrageenan is a non-toxic gelling agent safe in animals and humans as a potent HPV inhibitor. An anionic polymer derived from red algae, carrageenan has a long history of human use as a stabilizer and emulsifier in many industries. All three major classes of carrageenan act as extremely potent HPV inhibitors and block HPV infection by binding to the viral capsid, thus preventing attachment to the appropriate cell-surface heparan sulfate proteoglycans (HSPG) receptors.
- Control Gel: The intervention to be administered is:
  * a commercially available gel that does not contain carrageenan.
  * water-based, latex-condom compatible, clear, odourless, tasteless, and have similar viscosity as the carrageenan-containing gel.
  * also packaged in a similar plastic bottle with a disk cap that can be operated with one finger, and must be applied prior to anal intercourse during the entire study period. Around 15 ml of the personal lubricant will be dispensed into the hand and applied directly to the genital, anal, and condom surfaces prior to and as needed during anal sex. When sexual activity ceases, the water-based formulation of the gel allows it to be easily removed with lukewarm water.
  Control gel: A gel not containing carrageenan
Period: Overall Study
Arm/Group | Carrageenan-based Gel | Control Gel
Started | 127 | 128
Completed | 48 (Participants completed all 7 study visits.) | 51 (Participants completed all 7 study visits.)
Not Completed | 79 | 77

BASELINE CHARACTERISTICS:
Population: The description of baseline characteristics includes participants included in the interim analysis prior to trial termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carrageenan-based Gel | Control Gel | Total
Number analyzed (Participants) | 127 | 128 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] — The description of baseline characteristics includes participants included in the interim analysis prior to trial termination.
  years | 36.7 (14.2) | 37.0 (14.4) | 36.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 127 | 128 | 255
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  French Canadian | 48 | 50 | 98
  English Canadian | 17 | 20 | 37
  Latin American | 14 | 15 | 29
  European | 20 | 12 | 32
  Other | 28 | 31 | 59
Human immunodeficiency virus status, positive [Count of Participants; unit: Participants] | 33 | 35 | 68
HPV DNA status [Count of Participants; unit: Participants] — Anal samples were tested and typed for 36 different HPV types using the linear array assay from Roche. Participants were considered HPV positive if the anal sample was positive for any of the 36 different HPV types.
  Participants | 84 | 71 | 155

OUTCOME MEASURES:

1. Primary Outcome: Presence of a Newly Detected Anal Infection of a Specific HPV Type in a Man Who Was Negative for That HPV Type at Enrollment
Description: Detection of 36 different HPV types will allow for the assessment of new HPV types even among those already infected.
Time Frame: One year follow-up
Population: 201 participants were included in the intention to treat analyses. Of the 255 initially randomized, 45 were excluded because they only had one visit and 9 were excluded because HPV data was unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Carrageenan-based Gel | Control Gel
Number analyzed (Participants) | 98 | 103
Participants | 68 | 67

2. Secondary Outcome: Clearance of Anal Type-specific HPV Infections Found at Baseline
Description: Detection of 36 different HPV types will allow for the assessment of clearance of any HPV type or specific HPV types.
Time Frame: One year follow-up
Population: Of the 255 participants randomized at the time of interim analysis, there were 134 participants positive for HPV at baseline that had at least 2 visits with valid HPV results. These 134 participants were included in the clearance analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Carrageenan-based Gel | Control Gel
Number analyzed (Participants) | 68 | 66
Participants | 19 | 22

3. Secondary Outcome: Patient Adherence, Measured Via Questionnaires and Review of Patient Adverse Event Reports.
Description: Measured via questionnaires and review of patient adverse event reports. Adherence was defined as the number of times the gel was used during receptive anal intercourse divided by the number of receptive anal intercourse in the 7 days preceding each visit. Participants were considered adherent at a particular visit if they used the gel during receptive anal intercourse ≥ 50% of the time. This variable was analyzed at the visit level. Safety analyses are included in the adverse event reporting section.
Time Frame: One year follow-up
Population: Of the 255 participants randomized at the time of interim analysis, 210 participants had available follow-up and were included in adherence and safety analyses.
Measure: Count of Units; unit: visits
Units Other Than Participants: visits
Arm/Group | Carrageenan-based Gel | Control Gel
Number analyzed (Participants) | 127 | 128
Number analyzed (visits) | 428 | 441
visits | 361 | 389

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the participants follow-up (1 year).
Description: Adverse event (AE) data was collected from the weekly calendar, follow-up surveys, and nurses notes. Data from the weekly calendar and nurses notes included specific descriptions of the AE. AE data from the follow-up surveys was a yes no answer to the question of whether the participant experience any adverse events or adverse reactions.
Arm/Group | Carrageenan-based Gel | Control Gel
All-Cause Mortality (participants affected / at risk) | 0/102 | 1/108
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/108
Other Adverse Events (participants affected / at risk) | 61/102 | 43/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carrageenan-based Gel (N=102) | Control Gel (N=108)
Death (Infections and infestations) | 0 | 1 — Death, related to underlying HIV infection complicated by drug use.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Carrageenan-based Gel (N=102) | Control Gel (N=108)
Unusual pain during anal sex (Product Issues) | 4/75 (4) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Rectal bleeding in between anal sex (Product Issues) | 6/75 (6) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Unusual abdominal pain (Product Issues) | 2/75 (2) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Unusually painful defecation (Product Issues) | 0/75 (0) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Flatulence, constipation, urgency and/or fecal incontinence or diarrhea (Product Issues) | 0/75 (0) | 1/77 (1) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Rectal abscess/ulcer/fistulae (Product Issues) | 0/75 (0) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Anal discharge (Product Issues) | 2/75 (2) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Hemorrhoids (Product Issues) | 0/75 (0) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Itching, burning, edema or pain in the anorectal area (Product Issues) | 4/75 (4) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Anal fissures (Product Issues) | 0/75 (0) | 0/77 (0) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Other (Product Issues) | 3/75 (3) | 1/77 (1) — AE reported in calendar. Non-response for 27 in the carrageenan and 31 in the placebo arm.
Use of the gel caused discomfort/adverse reactions to you (Product Issues) | 18/99 (18) | 8/103 (8) — AE reported in survey. Non-response for 3 participants in the carrageenan and 5 in the placebo arm.
Use of the gel caused discomfort/adverse reactions to your partner(s) (Product Issues) | 13/99 (13) | 2/105 (2) — AE reported in survey. Non-response for 3 participants in the carrageenan and 5 in the placebo arm.
Reported bleeding following receptive anal intercourse (Product Issues) | 47/95 (47) | 43/101 (43) — AE reported in survey. Non-response for 7 participants in the carrageenan and 7 in the placebo arm.
Warts (Product Issues) | 6 (6) | 7 (7) — Conditions reported by nurse at the clinic visit.
Erythema (Product Issues) | 6 (6) | 9 (9) — Conditions reported by nurse at the clinic visit.
Abrasions (Product Issues) | 4 (4) | 2 (2) — Conditions reported by nurse at the clinic visit.
Inflammation (Product Issues) | 2 (2) | 0 (0) — Conditions reported by nurse at the clinic visit.
Fissures (Product Issues) | 3 (3) | 2 (2) — Conditions reported by nurse at the clinic visit.
Abscesses (Product Issues) | 1 (1) | 1 (1) — Conditions reported by nurse at the clinic visit.
Hemorrhoids (Product Issues) | 11 (11) | 7 (7) — Conditions reported by nurse at the clinic visit.
Venereal warts or condylomas (Product Issues) | 2/95 (2) | 3/92 (3) — Infections/conditions reported by participant in survey. Non-response for 7 participants in the carrageenan and 16 in the placebo arm.
Chlamydia (Product Issues) | 14 (14) | 12 (12) — Infections/conditions reported by participant in survey.
Lymphogranuloma vereneum (Product Issues) | 0 (0) | 1 (1) — Infections/conditions reported by participant in survey.
Anal or genital herpes (Product Issues) | 5 (5) | 5 (5) — Infections/conditions reported by participant in survey.
Syphilis (Product Issues) | 7 (7) | 7 (7) — Infections/conditions reported by participant in survey.
Gonorrhea (Product Issues) | 23 (23) | 10 (10) — Infections/conditions reported by participant in survey.
Ulcers or genital sores (Product Issues) | 0 (0) | 1 (1) — Infections/conditions reported by participant in survey.
Hepatitis B (Product Issues) | 0 (0) | 1 (1) — Infections/conditions reported by participant in survey.
Hepatitis C (Product Issues) | 0 (0) | 2 (2) — Infections/conditions reported by participant in survey.
HIV (Product Issues) | 1 (1) | 0 (0) — Infections/conditions reported by participant in survey.
Anal precancer (Product Issues) | 0 (0) | 1 (1) — Infections/conditions reported by participant in survey.
Cancer (Product Issues) | 0 (0) | 1 (1) — Infections/conditions reported by participant in survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02354144/Prot_SAP_000.pdf